CLINICAL TRIAL: NCT04640116
Title: Feasibility and Clinical Outcome of TIPS Combined With Subsequent Microwave Ablation in HCC Patients With Refractory Ascites
Brief Title: TIPS Combined With Microwave Ablation in HCC Patients With Refractory Ascites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZQFGF
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Liver Diseases; Portal Hypertension; Cirrhosis, Liver; Ascites; Hepatocellular Carcinoma
Keywords: Transjugular intrahepatic portosystemic shunt; refractory ascites; microwave ablation
MeSH Terms: conditions — Liver Diseases; Hypertension, Portal; Liver Cirrhosis; Ascites; Carcinoma, Hepatocellular | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIPS combined with microwave ablation (Experimental)
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt (TIPS); Procedure: microwave ablation (MWA)

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt (TIPS) — A needle punctured the portal vein through the transjugular approach. After a successful puncture, the parenchymal tract was dilated, and covered stents (GORE® VIATORR) were introduced. The specifications of the covered stents were 8 mm × 50 mm, 8 mm × 60 mm, 8 mm × 70 mm, and 8 mm × 80 mm. All of the diameters of the bare stents were 8 mm, and the lengths were 50-80 mm. The portal vein pressure was measured before and after shunt creation. After the insertion of TIPS, all of the patients received a diuretic treatment and a salt-limited diet until the ascites disappeared.
Procedure: microwave ablation (MWA) — MWA: After the patient's ascites disappears, MWA therapy will be performed. A MWA antenna was gradually inserted into the tumor along the predetermined angle under the guidance of Computed Tomography (CT). The whole thermal procedure was conducted under intravenous anesthesia. Vital signs were monitored during the procedure. The settings of the ablation parameters depended upon the manufacturer's recommendation and our experience. Ablation volume was determined by physicians according to liver function, tumor invasion site, and tumor stage. An upper abdominal CT scan was carried out immediately after the procedure to evaluate the ablation area and complications.

SUMMARY:
Transjugular intrahepatic portosystemic shunt (TIPS) could effectively decrease portal hypertension-related complications. This study intends to evaluate the efficacy and safety of TIPS combined with subsequent microwave ablation in HCC patients with refractory ascites.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) patients with refractory ascites (RA) have a very poor prognosis, and there are no effective treatments recommended by the guidelines. TIPS could downgrade the ascites and improve Child-Pugh scores. TIPS has been a common management model for RA for end-stage liver disease. There is no prospective study evaluating TIPS plus thermal ablation. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years
2. Diagnosis of HCC based on the European Association for the Study of the Liver
3. Tumor diameter ≤ 3cm
4. Refractory ascites based on International Ascites Club: (a) intensive diuretics (spironolactone 400 mg/d combined with furosemide 160 mg/d) and sodium-restricted diet (<90 mmoVd) for at least 1 week have no response; (b) lack of response to diuretic therapy; (c) early recurrence of ascites within 4 weeks; (d) Diuretic-induced complications. The grading of ascites was divided into mild ascites, moderate ascites, and large or gross ascites

Exclusion Criteria:

1. Congestive heart failure or severe valvular heart failure
2. Uncontrolled systemic infection or inflammation
3. Macroscopic vascular invasion or extrahepatic metastasis
4. Severe pulmonary hypertension
5. Severe renal insufficiency (except hepatogenic renal insufficiency) (6) rapidly progressive liver failure
6. Diffuse malignant liver tumor
7. Contrast agent allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 24 months
  the interval from TIPS to death or lost to follow-up

SECONDARY OUTCOMES:
change in Child-Pugh stage | 6 months
  the liver function stage change from C to B or from B to A
change in Child-Pugh scores | 6 months
  decrease of Child-pugh scores
Incidence of hepatic encephalopathy | 24 months
  the incidence of hepatic encephalopathy of patients accepting TIPS
Varices rebleeding rate | 24 months
  the incidence of varices bleeding of patients accepting TIPS

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Professor, Study Director — Second Affiliated Hospital of Guangzhou Medical University; Fei Gao, Professor, Study Director — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No